## **COVER PAGE**

STUDY TITLE: ASSESSMENT OF THREE BASIC PROGRESSIVE LENS DESIGNS

**REGISTRATION NUMBER:** NCT05252871

**DATE:** 09/27/2021

## **DATA ANALYSIS PLAN**

## **DATA ANALYSIS:**

Data analysis includes Analysis of Variance (ANOVA) or its non-parametric alternatives with post-hoc tests and correlation analysis:

- Repeated-measures ANOVA or its non-parametric alternatives are conducted since
  each participant experienced all three lens designs. This allows to assess the main
  effect of lens design while accounting for the repeated measures within participants.
  Influencing factors (age group, gender, previous lens design experience, lens power,
  add power) are included as independent variables to investigate their potential effects on
  the outcomes.
- Significant differences in the ANOVA or its non-parametric alternatives are further explored through post-hoc tests to determine which specific pairs of progressive lens designs (A, B, or C) or levels of influencing factors (age group, gender, previous lens design experience, lens power, add power) differ from each other.
- Correlation analyses are utilized to investigate the relationships between continuous variables (e.g., age) and the Likert scale responses.